CLINICAL TRIAL: NCT06221774
Title: An Open-Label, Multi-Cohort, Two-Stage, Phase Ib/II Clinical Study to Evaluate the Safety and Efficacy of TT-00420 Tablets Combined With Toripalimab Injection in Treating Advanced Urological Tumors
Brief Title: Safety and Efficacy of TT-00420 Tablets Combined With Toripalimab Injection in Advanced Urological Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-121
Record Dates: First submitted 2023-12-24; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Clear Cell Renal Carcinoma; Urothelial Carcinoma; Metastatic Castration-resistant Prostate Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase Ib: dose optimization phase (Experimental): Approximately 12 participants will be enrolled and randomized 1:1 into two different dosage groups:
  * Dose Group A (N=6): TT-00420 tablets 10mg QD + Toripalimab 240mg Q3W.
  * Dose Group B (N=6): TT-00420 tablets 8mg QD + Toripalimab 240mg Q3W.
  Interventions: Drug: TT-00420 + Toripalimab
- Phase II (Experimental): Based on the safety and efficacy data from Phase Ib, further cohorts will enroll participants with specific tumor types at the optimal dose of TT-00420 tablets:
  * Cohort 1 (N=10): Metastatic or unresectable advanced renal clear cell carcinoma (RCC).
  * Cohort 2 (N=10): Metastatic or unresectable advanced urothelial carcinoma (UC).
  * Cohort 3 (N=10): Metastatic castration-resistant prostate cancer (mCRPC).
  Interventions: Drug: TT-00420 + Toripalimab

INTERVENTIONS:
Drug: TT-00420 + Toripalimab — TT-00420 tablets in combination with Toripalimab injection

SUMMARY:
This Phase Ib/II clinical study is an open-label, multi-cohort, two-stage trial designed to assess the safety and efficacy of different doses of TT-00420 tablets in combination with Toripalimab injection for treating patients with advanced urological tumors. The study aims to evaluate the effectiveness of TT-00420 tablets at the optimal dose combined with Toripalimab in treating different types of advanced urological tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation, sign the informed consent with good compliance.
2. Age between 18-80 years.
3. ECOG performance status of 0 or 1; expected survival of at least 3 months.
4. Meeting all criteria for one of the following cancer types:

   * Renal Clear Cell Carcinoma:

     1. Pathologically and radiologically confirmed metastatic or unresectable advanced clear cell renal cell carcinoma.
     2. Failure after at least one systemic treatment for advanced or metastatic disease (including chemotherapy, targeted therapy, immunotherapy).
     3. At least one measurable lesion (RECIST 1.1).
   * Urothelial Carcinoma:

     1. Pathologically and radiologically confirmed metastatic or unresectable advanced urothelial carcinoma (including bladder, ureter, renal pelvis, and urethra).
     2. Failure or refusal to receive at least one systemic chemotherapy for advanced, recurrent/metastatic disease.
     3. Progression after one PD-1/PD-L1 inhibitor treatment.
     4. At least one measurable lesion (RECIST 1.1).
   * Prostate Cancer:

     1. Pathologically confirmed mCRPC with radiologically confirmed bone metastases or soft tissue metastases.
     2. Failure after at least one novel endocrine treatment for metastatic disease (including but not limited to abiraterone, enzalutamide).
     3. Failure or refusal of systemic chemotherapy.
     4. Baseline serum testosterone < 50 ng/dL (1.73 nmol/L).
     5. For participants without baseline soft tissue target lesions, baseline serum PSA ≥ 2 ng/mL and meeting PSA disease progression criteria per PCWG3.
5. Adequate major organ function, laboratory test criteria:

   * Hematology:

     1. Hemoglobin (HB) ≥ 90 g/L.
     2. Absolute Neutrophil Count (ANC) ≥ 1.5×109/L.
     3. Platelets (PLT) ≥ 75×109/L.
   * Biochemistry:

     1. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 × ULN (≤ 5 × ULN for liver/bone metastasis).
     2. Total Bilirubin (TBIL) ≤ 1.5 × ULN.
     3. Serum Creatinine ≤ 1.5×ULN or Creatinine Clearance ≥ 30 mL/min.
   * Coagulation:

   Activated Partial Thromboplastin Time (APTT), International Normalized Ratio (INR), Prothrombin Time (PT) ≤ 1.5×ULN.
6. Fertile women must agree to contraception during the study and for 3 months after the last administration of the study drug.

[Failure Definition: Disease progression during treatment or after the last treatment, or intolerable toxicity due to side effects during treatment. Prior neoadjuvant or adjuvant treatment is allowed. If disease relapse or progression occurs within 6 months after the end of neoadjuvant/adjuvant treatment, it is considered a failure of first-line treatment for progressive disease.]

Exclusion Criteria:

1. Primary pure neuroendocrine cancer (except post-treatment neuroendocrine differentiation).

2. Other antitumor treatments within 4 weeks or 5 half-lives (whichever is shorter) before the start of the study treatment (except androgen deprivation therapy for prostate cancer patients, such as LHRH agonists or antagonists, bicalutamide, flutamide, etc.), or not yet recover from the toxicity of previous treatments (except ≤ G1 adverse events or tolerable G2 alopecia, fatigue/asthenia, and neuropathy caused by trauma at baseline).

3. Concurrent diseases/history:

1. Clinically significant hemoptysis (> 50 mL per day) within 3 months before enrollment; significant clinical bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcers, baseline fecal occult blood and above.
2. Arteriovenous thrombotic events within 6 months before enrollment, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis (except venous thrombosis caused by previous chemotherapy with venous catheterization judged by the investigator as cured), and pulmonary embolism.
3. Hypertension not well controlled with stable dose antihypertensive treatment (systolic pressure > 150 mmHg or diastolic pressure > 100 mmHg); myocardial infarction, severe/unstable angina, NYHA class 2 or above heart failure, clinically significant supraventricular or ventricular arrhythmias, prolonged QT interval, and symptomatic congestive heart failure within 6 months before baseline/screening.
4. Interstitial lung disease, non-infectious pneumonia, and other non-specific pneumonias (e.g., pulmonary fibrosis, interstitial pneumonia).
5. Active infection requiring antibiotic treatment within 4 weeks before the first administration of the study drug, or unexplained fever > 38.5°C during screening or before the first administration of the study drug (fever due to tumor reasons judged by the investigator is allowed for enrollment); active tuberculosis.
6. Live attenuated vaccine vaccination history within 28 days before the first study drug administration or expected live attenuated vaccine vaccination during the study (including COVID-19 vaccine).
7. HIV infection or known acquired immunodeficiency syndrome (AIDS).
8. Active HBV infection (other abnormal HBV serology tests besides hepatitis B surface antibody positive or ≥ ULN, HBV DNA copy number required to confirm activity) and/or HCV infection (HCV RNA copy number required to confirm activity if hepatitis C virus antibody is abnormal).
9. Major surgery, extensive radiotherapy within 28 days before enrollment, or local palliative radiotherapy within 2 weeks.
10. Baseline: ≥ G2 peripheral neuropathy; active brain metastases, carcinomatous meningitis, spinal cord compression, or imaging studies (CT or MRI) at screening showing brain or leptomeningeal disease (patients with brain metastases who have completed treatment and stabilized symptoms within 14 days before enrollment are allowed, but must be evaluated by cranial MRI, CT, or venography to confirm no symptoms of cerebral hemorrhage).
11. Factors significantly affecting oral drug absorption, such as inability to swallow, history of total gastrectomy, short bowel syndrome, or clinically significant intestinal obstruction.
12. Participants who have received or are preparing to receive allogeneic bone marrow transplantation or organ transplantation.
13. History of severe allergy, immunostress, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins; hypersensitivity or allergy to any component of Toripalimab injection.
14. Active autoimmune diseases requiring systemic treatment within 2 years before the first administration of the study drug. Replacement therapy is not considered systemic treatment.
15. Diagnosed with immunodeficiency or receiving systemic corticosteroid treatment or any form of immunosuppressive therapy, and continuing to use within 2 weeks before the first administration of the study drug.

4. Pregnant, breastfeeding, or planning to become pregnant during the study. 5. Other serious physical or mental illnesses or laboratory test abnormalities that may increase the risk of participating in the study, interfere with study results, or patients deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Treatment-Related Adverse Events [Safety and Tolerability] in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  To assess the incidence of adverse events at different doses of TT-00420 tablets combined with Toripalimab Injection.
Types of Treatment-Emergent Adverse Events and Treatment-Related Adverse Events [Safety and Tolerability] in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  To assess the types of adverse events at different doses of TT-00420 tablets combined with Toripalimab Injection.
Severity of Treatment-Emergent Adverse Events and Treatment-Related Adverse Events [Safety and Tolerability] in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  To assess the severity of adverse events at different doses of TT-00420 tablets combined with Toripalimab Injection per CTCAE V5.0.
ORR in Phase II | Through study of Phase II, an average of 1 year
  Objective Response Rate (ORR) according to RECIST v1.1 for renal cell carcinoma, urothelial carcinoma, and prostate cancer (with baseline target lesions).
PSA Response Rate in Phase II | Through study of Phase II, an average of 1 year
  PSA Response Rate (including PSA50 and PSA30, per PCWG3) for prostate cancer.

SECONDARY OUTCOMES:
ORR in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  Objective Response Rate (ORR) according to RECIST v1.1 for renal cell carcinoma, urothelial carcinoma, and prostate cancer (with baseline target lesions).
PSA Response Rate in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  PSA Response Rate (PCWG3 for prostate cancer)
DCR in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  Disease Control Rate (DCR)
PFS in months in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  Progression-Free Survival (PFS)
OS in months in Phase Ib | Through study of Phase Ib, an average of 12 weeks
  Overall Survival (OS)
DCR in Phase II | Through study of Phase II, an average of 1 year
  Disease Control Rate (DCR)
PFS in months in Phase II | Through study of Phase II, an average of 1 year
  Progression-Free Survival (PFS)
OS in months in Phase II | Through study of Phase II, an average of 1 year
  Overall Survival (OS)
Incidence of Treatment-Emergent Adverse Events and Treatment-Related Adverse Events [Safety and Tolerability] in Phase II | Through study of Phase II, an average of 1 year
  To assess the incidence of adverse events at different doses of TT-00420 tablets combined with Toripalimab Injection.
Types of Treatment-Emergent Adverse Events and Treatment-Related Adverse Events [Safety and Tolerability] in Phase II | Through study of Phase II, an average of 1 year
  To assess the types of adverse events at different doses of TT-00420 tablets combined with Toripalimab Injection.
Severity of Treatment-Emergent Adverse Events and Treatment-Related Adverse Events [Safety and Tolerability] in Phase II | Through study of Phase II, an average of 1 year
  To assess the severity of adverse events at different doses of TT-00420 tablets combined with Toripalimab Injection per CTCAE V5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China